CLINICAL TRIAL: NCT00123526
Title: Active Living and Healthy Diet at the Workplace
Brief Title: Workplace-Sponsored Diet and Exercise Program to Reduce Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Stephenie Lemon, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 223; R01HL079483 (NIH)
Record Dates: First submitted 2005-07-21; First posted 2005-07-25 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Heart Diseases | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Worksite intervention
  Interventions: Behavioral: Diet; Behavioral: Physical Activity
- 2 (No Intervention): Receive no intervention

INTERVENTIONS:
Behavioral: Diet — Participants will also follow a healthy diet, characterized by higher intakes of fruits, vegetables, fish, poultry, legumes, and whole grains. Participants will consume less high fat foods and refined grains, and reduce their total caloric intake through smaller portion sizes.
  Arms: 1
Behavioral: Physical Activity — The intervention will promote active living, in which physical activity is incorporated into each participants' daily routine.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of an environmental worksite intervention to reduce obesity among hospital employees.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity is a significant public health problem in the United States, prompting policy makers and researchers to call for action against the epidemic. Obesity and associated health conditions affect all age groups and both genders, yet disproportionately affect racial and ethnic minorities. Health consequences of obesity include high blood pressure, high cholesterol, hyperinsulinemia, type 2 diabetes, heart disease, stroke, gallbladder disease, arthritis, sleep disturbances, breathing problems, and certain types of cancer. Hospitals are important worksite environments that employ large numbers of people in diverse job categories from diverse educational and socioeconomic backgrounds.

DESIGN NARRATIVE:

The purpose of this study is to promote weight loss among those who are overweight and obese, and prevent weight gain among those of normal weight through an environmental intervention targeted to all employees at six hospitals in central Massachusetts. The hospitals will be matched according to size, and within each matched pair randomly assigned to either the intervention or control group. The intervention will promote active living, in which physical activity is incorporated into each participants' daily routine. Participants will also follow a healthy diet, characterized by higher intakes of fruits, vegetables, fish, poultry, legumes, and whole grains. Participants will consume less high fat foods and refined grains, and reduce their total caloric intake through smaller portion sizes.

ELIGIBILITY:
Inclusion criteria:

* Works at least 20 hours per week at a participating hospital
* Speaks English or Spanish

Exclusion criteria:

* Works at only one hospital within the participating hospital system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 899 (Actual)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Body mass index | Measured at Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Stephenie Lemon, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States